CLINICAL TRIAL: NCT07406152
Title: Efficacy and Safety of ZKARE® Gel and Its Accessory ZKAPI® in the Treatment of Chronic Ulcers: a Prospective, Randomized, Controlled Clinical Investigation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Bioaraba Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZKARE-PIC01-2025
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Ulcers
Keywords: Pressure ulcers; Hyaluronic acid; Wound healing; Topical gel; venous leg ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZKARE® (Experimental): Participants assigned to this arm receive standard wound care plus topical application of the investigational gel ZKARE®, applied using the ZKAPI® applicator during each wound-care session.
  Interventions: Device: ZKARE®
- Standard Wound Care (Active Comparator): Participants assigned to this arm receive standard wound management according to routine clinical practice, without the use of the investigational product.
  Interventions: Procedure: Standard Wound Care

INTERVENTIONS:
Device: ZKARE® — ZKARE® is applied topically after routine wound cleansing and debridement. Using the sterile ZKAPI® applicator, the gel is distributed to fully cover the wound bed, including irregular or cavitated areas. The treated wound is then covered with the appropriate secondary dressing following standard clinical practice. The application is repeated at each treatment session until complete closure or the end of the 12-week follow-up period. All sessions include RESVECH 2.0 scoring, standardized photographs, and safety assessments
  Arms: ZKARE®
Procedure: Standard Wound Care — Standard care includes wound cleansing, debridement when required, and selection of secondary dressings according to wound characteristics such as exudate level, infection status, depth, and perilesional skin condition. No investigational gel is applied. At each treatment visit and follow-up time point, standardized wound photographs, RESVECH 2.0 scoring, closure metrics, and safety assessments are recorded according to the same schedule as the investigational arm.
  Arms: Standard Wound Care

SUMMARY:
This prospective, randomized, single-blind, controlled clinical investigation evaluates the efficacy and safety of ZKARE®, a topical polymeric gel dressing, and its accessory applicator ZKAPI®, for the treatment of chronic, hard-to-heal ulcers. The study includes 134 ulcers of different etiologies-pressure ulcers, neuropathic diabetic foot ulcers, and venous leg ulcers-meeting predefined selection criteria. Participants are randomized to receive either ZKARE® in addition to standard wound care or standard care alone.

The primary efficacy endpoint is the change in wound condition assessed through the RESVECH 2.0 scale, recorded at baseline and throughout treatment and follow-up visits. The primary safety endpoint is the incidence of serious adverse events (SAEs). Secondary outcomes include percentage and rate of wound closure, total closure rate, estimated time to full closure, quality-of-life measures (DLQI), patient satisfaction, investigator global assessment, cost-effectiveness, and product usability. The study aims to generate evidence on the performance, safety, and clinical usefulness of ZKARE® for chronic wound management.

DETAILED DESCRIPTION:
Chronic ulcers such as pressure ulcers, neuropathic diabetic foot ulcers and venous leg ulcers frequently fail to follow normal healing phases and require comprehensive management. Many existing dressings act through a single mechanism and are limited in effectiveness for complex or exudative wounds. ZKARE® is a sterile, biocompatible polymeric gel intended for topical use that provides a moist microenvironment, absorbs excess exudate and contributes to bacterial control. The product is applied using ZKAPI®, a sterile Luer-Lock applicator designed to improve precision and ease of administration.

This prospective, randomized, single-blind, controlled clinical investigation compares ZKARE® plus standard care with standard care alone in 134 chronic ulcers of different etiologies. Patients may contribute more than one ulcer if lesions are independent. After informed consent, ulcers are randomized, and treatment sessions follow routine clinical practice, with ZKARE® added only in the investigational arm. Blinding is maintained by preventing direct visualization of the wound and through iso-appearance of materials. Follow-up visits occur at approximately 2, 4, 8 and 12 weeks.

The primary efficacy endpoint is the change in RESVECH 2.0 score, recorded at baseline, each treatment session and all follow-up visits; a ≥2-point improvement at Week 4 is considered clinically relevant. The primary safety endpoint is the incidence of serious adverse events. Secondary outcomes include percentage and rate of wound closure, total closure rate, estimated time to full closure, DLQI, patient satisfaction, investigator global assessment, usability and cost-effectiveness, as well as non-serious adverse events.

Group comparisons use appropriate statistical tests for categorical and continuous variables, repeated-measures analyses and ANCOVA where applicable, under an intention-to-treat approach. The sample size of 134 ulcers gives 80% power to detect expected differences in RESVECH 2.0 change. The study aims to evaluate the clinical performance and safety of ZKARE® and ZKAPI® in the treatment of chronic hard-to-heal ulcers

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years).
* Presence of at least one chronic hard-to-heal ulcer, including any of the following etiologies: Grade II, III or IV pressure ulcers; neuropathic diabetic foot ulcers (grade I, II or III), Wagner Grade I-III or Texas 0, I, II, III / Stage B; class C6/C6r venous leg ulcers measured with CEAP scale ; neuro-ischaemic ulcers with adequate distal perfusion (ABI/ITB ≥ 0.7-0.89; mild PAD); mixed-etiology venous ulcers and any chronic lower-limb lesion with palpable distal pulses.
* Ulcer size between 1 cm² and 100 cm².
* Ability and willingness to comply with all study visits and procedures according to the clinical protocol.
* Ability to understand and sign the informed consent, obtained before performing any protocol-specific procedures.

Exclusion Criteria:

* Ulcers of etiologies not listed in the inclusion criteria.
* Ischaemic, neoplastic or atypical ulcers.
* Severe comorbidities judged to compromise safety or study compliance, including: severe malnutrition, palliative/terminal status, severe anemia, decompensated heart failure, chronic kidney disease stage III/IV or in dialysis.
* Ulcers with moderate-severe or severe infection per PEDIS-IDSA infection grading scale.
* Known allergy or sensitivity to any component of the investigational product.
* Any condition that, in the investigator's opinion, may compromise patient safety or adherence to the protocol.
* Pregnancy or planned breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
RESVECH Scale 2.0 | 12 weeks or wound healing
  Change in the RESVECH 2.0 wound assessment scale, which evaluates wound size, depth, granulation tissue quality, exudate amount/type, clinical signs of infection/inflammation, and perilesional skin condition.
  Measured at baseline and at each treatment and follow-up visit until complete closure or at week 12. A ≥2-point improvement at week 4 is considered clinically relevant.
Incidence of Serious Adverse Events (SAEs) | 12 weeks
  Incidence, frequency, and nature of serious adverse events during the study.

SECONDARY OUTCOMES:
Wound Closure Rate (mm²/day) | 12 weeks
  Rate of epithelialization based on the area healed divided by the time since treatment initiation.
  Assessed at each treatment and follow-up visit.
Percentage of Wound Closure (%) | 12 weeks
  Percentage reduction of the initial wound area at each assessment. A ≥30% reduction by week 4 is considered clinically relevant.
  Kaplan-Meier curves may be used to evaluate closure thresholds (≥30%-90%).
Total Wound Closure (%) | 12 weeks
  Percentage of wounds achieving complete epithelialization.
Estimated Time to Full Closure (days) | 12 weeks
  For wounds not completely healed by week 12, linear regression based on closure rate is used to estimate time to complete healing.
Cost-Effectiveness Analysis (Healthcare Resources Used) | 12 weeks
  Quantification of materials, products, consumables, and healthcare professional time in each treatment session.
  Reported as €/patient.
Dermatology Life Quality Index (DLQI) Score | 12 weeks
  Change in DLQI score (0-30), with higher scores indicating worse dermatology-related quality of life.
Patient Satisfaction (Likert Scale) | 12 weeks
  Patient satisfaction rated at study end (Very dissatisfied, dissatisfied, neutral, satisfied and very satisfied).
  Outcome to be reported as the percentage of "Satisfied" + "Very satisfied" answers.
Investigator Global Assessment (IGA) | 12 weeks
  Clinical impression of overall wound evolution (Worsening / No improvement / Mild improvement / Significant improvement).
  Outcome to be reported as the percentage of mild or significant improvement achievement.
Incidence of Non-Serious Adverse Events (AEs) | 12 weeks
  Recording of the incidence and nature of all non-serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Álava, Spain

IPD SHARING:
Plan to Share IPD: No